CLINICAL TRIAL: NCT01352962
Title: A Phase I Study of Gemcitabine, Carboplatin and Lenalidomide (GCL) for Treatment of Patients With Advanced/Metastatic Urothelial Carcinoma (UC) and Other Solid Tumors
Brief Title: Gemcitabine, Carboplatin, and Lenalidomide for Treatment of Advanced/Metastatic Urothelial Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 110140; 11-C-0140
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-09-15

CONDITIONS: Urethral Neoplasms; Neoplasms, Urethral; Cancer of the Urethra; Urethral Cancer
Keywords: Dose Limiting Toxicity; Urethra Cancer; Carcinoma of the Bladder; Cancer of the Renal Pelvis; Ureter Cancer; Urethral Cancer; Solid Tumor; Pancreatic Cancer; Ovarian Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Urethral Neoplasms; Urinary Bladder Neoplasms; Ureteral Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Standard of Care plus escalating doses of Lenalidomide
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Lenalidomide
- Arm 2 (Experimental): Lenalidomide Lead for 14 days + standard of care + lenalidomide MTD
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Lenalidomide

INTERVENTIONS:
Drug: Gemcitabine — 1,000mg/m2 IVPB over 30 min x 1
Drug: Carboplatin — AUC 5** IVPB over 30 min x 1
Drug: Lenalidomide — Escalating Doses starting at 2.5 po daily up to 25 mg po daily until MTD is reached.

SUMMARY:
Background:

- Gemcitabine and carboplatin are chemotherapy drugs used to treat several types of cancer, including cancer of the pancreas, bladder, ovaries, and lung. Lenalidomide, a drug that prevents the growth of new blood vessels in tumors, has been approved for treatment of certain blood cancers, but it has not yet been approved for use in combination with gemcitabine and carboplatin. Researchers are interested in determining the safest and most effective dose of this combined form of chemotherapy for solid tumors, particularly for urothelial cancer (tumors of the bladder, urethra, ureter, or renal pelvis).

Objectives:

* To evaluate the safety and effectiveness of combined lenalidomide, gemcitabine, and carboplatin as a treatment for solid tumor cancers.
* To evaluate the safety and effectiveness of combined lenalidomide, gemcitabine, and carboplatin as a treatment for urothelial (bladder) cancer.

Eligibility:

* Individuals at least 18 years of age who have been diagnosed with solid tumors that have not responded to standard treatments.
* Individuals at least 18 years of age who have been diagnosed with urothelial cancer that has not responded to standard treatments.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and tumor imaging studies.
* Participants with urothelial cancer will receive lenalidomide alone for the first 14 days of a 21-day cycle before starting the first full treatment cycle.
* All participants will receive gemcitabine on days 1 and 8, and carboplatin on day 1 only, of every 21-day treatment cycle. Lenalidomide will be taken daily at home for the first 14 days of each cycle. Participants will be asked to take aspirin or other medications to prevent the possibility of blood clots.
* Participants may receive up to six cycles of treatment with this combination. If after six cycles the cancer has not grown or has shrunk, participants may continue to take lenalidomide alone for an additional 6 months (total of 12 months of therapy) or until the cancer recurs.
* Participants will be monitored with blood samples, physical examinations, and tumor imaging studies through the cycles of treatment.
* After the end of the last treatment cycle, participants will have followup visits every 3 months for the next 18 months, then every 6 months for another 18 months, and then yearly.

DETAILED DESCRIPTION:
BACKGROUND:

* Gemcitabine plus carboplatin is an accepted first-line therapy in patients unfit for cisplatin chemotherapy with metastatic urothelial carcinoma or other solid tumor malignancies.
* Both non-clinical and clinical data support targeting angiogenesis in urothelial carcinoma and other solid tumors.
* Both non-clinical and clinical data support targeting the immune system in urothelial carcinoma and other solid tumors.
* Lenalidomide has both anti-angiogenic and potent immunomodulatory properties.
* Lenalidomide has been safely coadministered with cytotoxic therapy in patients with solid tumors and non-clinical studies demonstrate possible synergy with gemcitabine.

OBJECTIVES:

Primary

- To establish the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of lenalidomide which can be safely combined with gemcitabine and carboplatin in patients with advanced/metastatic UC and other solid tumors that are unfit for cisplatin.

Secondary

* To preliminarily evaluate the progression free survival, response rate and overall survival in patients with advanced/metastatic UC and other solid tumors treated with the combination of lenalidomide, gemcitabine, and carboplatin.
* To determine the effects of treatment on a set of 4 laboratory parameters (including Treg, sIL-2R, VEGF and CTC.) in the expansion cohort of patients with bladder cancer treated at the MTD.

ELIGIBILITY:

* Adult patients with histologic documentation of an advanced solid tumor with unresectable or metastatic disease.
* Urothelial cancer patients should be ineligible for cisplatin based on one or more of the following:
* Calculated creatinine clearance of < 60 mL/min (but greater than or equal to 30 mL/min)
* Solitary kidney
* Karnofsky Performance Status < 80%
* No prior combination systemic chemotherapy for metastatic disease allowed for patients with UC, except single agent radiosensitizing chemotherapy (not considered prior systemic therapy), or prior neoadjuvant or adjuvant systemic chemotherapy (including cisplatin-based) is allowed provided if it was completed (Bullet) 6 months prior to diagnosis of metastatic disease; or prior intravesical therapy is permitted. Up to 1 line of chemotherapy in the metastatic setting is permitted for non UC patients.
* Laboratory evaluation must meet safety requirements, including a creatinine clearance greater than 30 using the Cockroft-Gault formula; may not be pregnant or breast-feeding.

DESIGN:

* This is a single-institution phase I study of gemcitabine (1000 mg/m2 on days 1 and 8) and carboplatin (AUC 5 on day 1) plus escalating doses of lenalidomide (GCL) in patients with advanced/metastatic UC and other solid tumors ineligible for cisplatin therapy. Lenalidomide will be administered once daily on days 1 through 14 every 21 days at escalating dose. An expansion cohort at the MTD of an additional 15 patients with bladder cancer will be enrolled in order to determine whether there are differences between pre-treatment and post-treatment levels of the following parameters: Treg, sIL- 2R, VEGF and CTC.
* Patients will receive a total of 6 cycles of gemcitabine and carboplatin in combination with lenalidomide unless disease progression or unacceptable toxicity occurs. Patients who achieve stable disease, a partial response, or a complete response after completion of 6 cycles will be eligible to continue lenalidomide alone at the same dose and schedule until disease progression. Restaging evaluations will occur after every 3 cycles of treatment (approximately 9 weeks).
* Based on a standard 3+3 design with 4 dose levels per cohort, a maximum of 24 patients, with the potential for an additional 3 patients with CrCl>60 mL/min, may need to be evaluated to determine the dose limiting toxicities (DLTs) and maximum tolerated dose (MTD) of lenalidomide in this combination therapy. With an expansion cohort of 15 patients at MTD, a total of 42 subjects may be enrolled over 1.5 -3 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Dose Escalation cohort only

- Adult patients with histologic documentation of an advanced solid tumor for whom gemcitabine and carboplatin would be appropriate first line therapy, including but not limited to urothelial cancer, non-small cell lung cancer, pancreatic and ovarian carcinoma.

Expansion cohort only

Patients must have a histologically confirmed diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis. Confirmation may be obtained from any CLIA certified lab.

OR

-Patient must have a histologically confirmed diagnosis of non-transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis including but not limited to squamous cell, neuroendocrine, adenocarcinoma including urachal and sarcomatoid. Confirmation may be obtained from any CLIA certified lab.

All patients

* Unresectable or metastatic disease
* Urothelial cancer patients should be ineligible for cisplatin based on one or more of the following:
* Calculated creatinine clearance of < 60 mL/min (but greater than or equal to 30 mL/min)
* Solitary kidney
* Karnofsky Performance Status < 80%
* Age greater than or equal to 18 years of age; UC is not a common cancer in children and without proven benefit, this combination of chemotherapy agents presents too great a risk for conducting as a phase I study in children.
* Karnofsky Performance Status greater than or equal to 60%
* Required Initial Laboratory Values:
* Absolute neutrophil count greater than or equal to 1.2 x 10(9)/L
* Platelets greater than or equal to 100 x 10(9)/L
* Bilirubin less than or equal to 1.5 times the upper limit of normal for the institution or less than or equal to 3 mg/dl in a subject with Gilbert Syndrome
* Aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 3 times the ULN for the institution (less than or equal to 5 times the ULN is acceptable if liver has tumor involvement).
* Serum creatinine < 2 or calculated creatinine clearance (CrCl) greater than or equal to 30 mL/min
* Ability to understand and willingness to sign the written informed consent document.
* Patients must be able to swallow whole capsules. Capsules must not be crushed or chewed; capsules must not be opened.

EXCLUSION CRITERIA:

* For urothelial cancer patients, no prior combination systemic chemotherapy for metastatic disease, except:
* Single-agent radiosensitizing chemotherapy is not considered prior systemic therapy
* Prior neoadjuvant or adjuvant systemic chemotherapy (including cisplatin-based) is allowed provided it was completed greater than or equal to 6 months prior to the diagnosis of metastatic disease
* Prior intravesical therapy is permitted
* For non-urothelial cancer patients, no more than 1 prior line of combination systemic chemotherapy for metastatic disease is allowed
* Less than or equal to 2 weeks since radiation therapy
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy. Patients that are on anticoagulation therapy for DVT will be allowed to enroll and continue on the treatment dose of enoxaparin or other anticoagulation such a warfarin.
* Patients with contraindications to anticoagulation therapy for deep venous thrombosis such as:
* Patients on full treatment dose of anticoagulation such as those patients being treated for a deep vein thrombosis or pulmonary embolus.
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1
* Anticipation of need for major surgical procedure during the course of the study

Those patients that develop DVTs during the study will be treated with anticoagulants and in certain cases, will continue on the protocol.

* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 14 days and again within 24 hours prior to starting Cycle 1 of lenalidomide. Further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy. A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Inability to comply with study and/or follow-up procedures
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide, gemcitabine or carboplatin, or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Due to the possibility of infection reactivation, patients who are known seropositive for or who have active viral infection with human immunodeficiency virus (HIV) are NOT eligible.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09-26 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
dose limiting toxicity (DLT) | Maximum Tolerated Dose (MTD)
  any grade 3 or 4 toxicity with exceptions listed in protocol; MTD is one dose level below the dose that induces DLT in more than 1/6 patients

SECONDARY OUTCOMES:
response rate | every 3 months for the first 18 months, every 6 months for the subsequent 18 months, then yearly
  Percentage of patients whose cancer shrinks or disappears after treatment
progression free survival | every 3 months for the first 18 months, every 6 months for the subsequent 18 months, then yearly
  time during which a patient shows no signs or symptoms of the growth or the spreading of a tumor
overall survival | every 3 months for the first 18 months, every 6 months for the subsequent 18 months, then yearly
  The length of time from the start of treatment that patients are still alive
effects of treatment on Treg, sIL-2R, VEGF, CTC and CEC | baseline, lead-in day 8, lead-in day 14 and C1D8
  determine the effects of treatment on a set of 5 laboratory parameters (including Treg, sIL-2R, VEGF, CTC and CEC in the expansion cohort of patients with bladder cancer treated at the MTD

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI

REFERENCES:
- [Background] Dredge K, Horsfall R, Robinson SP, Zhang LH, Lu L, Tang Y, Shirley MA, Muller G, Schafer P, Stirling D, Dalgleish AG, Bartlett JB. Orally administered lenalidomide (CC-5013) is anti-angiogenic in vivo and inhibits endothelial cell migration and Akt phosphorylation in vitro. Microvasc Res. 2005 Jan;69(1-2):56-63. doi: 10.1016/j.mvr.2005.01.002. PMID 15797261
- [Background] Corral LG, Haslett PA, Muller GW, Chen R, Wong LM, Ocampo CJ, Patterson RT, Stirling DI, Kaplan G. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. J Immunol. 1999 Jul 1;163(1):380-6. PMID 10384139
- [Background] Schafer PH, Gandhi AK, Loveland MA, Chen RS, Man HW, Schnetkamp PP, Wolbring G, Govinda S, Corral LG, Payvandi F, Muller GW, Stirling DI. Enhancement of cytokine production and AP-1 transcriptional activity in T cells by thalidomide-related immunomodulatory drugs. J Pharmacol Exp Ther. 2003 Jun;305(3):1222-32. doi: 10.1124/jpet.102.048496. Epub 2003 Mar 20. PMID 12649301
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0140.html